CLINICAL TRIAL: NCT02825277
Title: Utero-placental Vascularisation in Normal and Preeclamptic and Intra-uterine Growth Restriction Pregnancies: Third Trimester Quantification Using 3D Power Doppler With Comparison to Placental Vascular Morphology
Brief Title: Utero-placental Vascularisation in Normal and Preeclamptic and Intra-uterine Growth Restriction Pregnancies
Acronym: EVUPA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2013-A01049-36
Record Dates: First submitted 2016-06-30; First posted 2016-07-07 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-07

CONDITIONS: Preeclampsia; Intra-uterine Growth Restriction
Keywords: 3D Power Doppler; uteroplacental vascularization; preeclampsia; intra-uterine growth restriction; placental morphology
MeSH Terms: conditions — Pre-Eclampsia | interventions — Echocardiography, Doppler

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pathological group (Other): pregnant women with preeclampsia and/or IUGR pregnancy with a planned or semi-urgent caesarean section or vaginal delivery will be recruited into this study.
  Interventions: Device: Doppler
- physiological group (Other): pregnant women with normal pregnancy with a planned caesarean section or vaginal delivery will be recruited into this study
  Interventions: Device: Doppler

INTERVENTIONS:
Device: Doppler — acquisition of 3D power Doppler of uteroplacental vascularization unit in 72h before delivery and morphological analysis for placenta

SUMMARY:
Introduction

Preeclampsia (PE) and intra-uterine growth restriction (IUGR) are two major pregnancy complications related to chronic utero-placental hypoperfusion. Three-dimensional power Doppler (3DPD) angiography has been used for the evaluation of utero-placental vascularisation and three vascular indices have been calculated: the vascularisation index (VI), flow index (FI) and vascularisation-FI (VFI). However, several technical endpoints hinder the clinical use of 3DPD as physical characteristics and machine settings may affect 3DPD indices, and so its clinical significance is not yet clear.

Objectives

The primary objective is to better understand the clinical significance of 3DPD indices by evaluating the relationship between these indices and placental morphometry. Secondary objectives are (i) to determine the impact of machine settings and physical characteristics on 3DPD indices, and (ii) to evaluate physio-pathological placental vascularisation patterns.

Methods and analysis

This is a prospective controlled study. We expect to include 112 women: 84 with normal pregnancies and 28 with PE and/or IUGR (based on our former cohort study on 3DPD indices for PE and/or IUGR prediction (unpublished data)). Within 72 h before planned or semi-urgent caesarean section, utero-placental 3DPD images with five different machine settings will be acquired. Placentas will be collected and examined after surgery and stereological indices (volume density, surface density, length density) calculated. The 3DPD indices (VI, FI and VFI) of the placenta and adjacent myometrium will be calculated. Correlation between Doppler and morphological indices will be evaluated by Pearson or Spearman tests. Agreement between 3DPD indices and morphological indices will be assessed by Bland and Altman plots. The impact of Doppler settings and maternal characteristics on 3DPD indices will be evaluated with a multivariate linear regression model.

ELIGIBILITY:
General Inclusion Criteria:

* Age ≥18 years and ≤65 years Fetal anomalies
* Gestational age ≥30 gestational weeks
* With social insurance
* With written consent for participation
* With medical examination

Physiological group Inclusion Criteria

* Hospitalised pregnant women with scheduled or semi-urgent caesarean section according to national HAS recommendations or Hospitalised pregnant women with scheduled vaginal delivery.
* Normal pregnancy issues
* Normal fetal morphology

Pathological group Inclusion Criteria

* Pregnant women with preeclampsia and/or IUGR pregnancy
* Hospitalised pregnant women with scheduled or semi-urgent caesarean section or hospitalised pregnant women with scheduled vaginal delivery.

Exclusion Criteria:

* Fetal morphological abnormalities that may influence fetal circulation
* Maternal or fetal vital urgency
* Multiple pregnancy
* Non-placental origin IUGR
* Language barrier
* Patient under legal protection

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2013-12; Primary Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Measure of 3D power Doppler indice : the vascularization index (VI) | through study completion, an average of 42 month
Measure of 3D power Doppler indice : blood flow (the flow index (FI) | through study completion, an average of 42 month
Measure of of 3D power Doppler indice : the vascularization-flow index (VFI) | through study completion, an average of 42 month
Measure of volume density (morphological analysis) | through study completion, an average of 42 month
Measure of surface density (morphological analysis) | through study completion, an average of 42 month

CONTACTS AND LOCATIONS:
Overall Officials: Olivier MOREL, MD, PhD, Principal Investigator — Inserm U947, IADI, Nancy, France
Locations (1):
- Pr Olivier MOREL, Vandœuvre-lès-Nancy, France

REFERENCES:
- [Background] Duan J, Chabot-Lecoanet AC, Perdriolle-Galet E, Christov C, Hossu G, Cherifi A, Morel O. Utero-placental vascularisation in normal and preeclamptic and intra-uterine growth restriction pregnancies: third trimester quantification using 3D power Doppler with comparison to placental vascular morphology (EVUPA): a prospective controlled study. BMJ Open. 2016 Mar 31;6(3):e009909. doi: 10.1136/bmjopen-2015-009909. PMID 27033959